CLINICAL TRIAL: NCT04784208
Title: A Study to Determine the Validity and Sensitivity of 'Questionnaire to Screen for HYpothyroidism' (Q'SHY)
Acronym: STRI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Abbott (Industry)
Responsible Party: Sponsor
Other Study IDs: EPIDI077
Record Dates: First submitted 2021-02-25; First posted 2021-03-05 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Hypothyroidism; Healthy
MeSH Terms: conditions — Hypothyroidism | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Arm 1-Healthy Volunteers: Arm 1: Subjects from the general population who are naïve to their hypothyroid status.
  The Subjects will be randomly selected and will be equally stratified between genders and socio-economics statuses from places where groups of general populations are located
  Interventions: Diagnostic Test: Blood test for Thyroid stimulating hormone (TSH)
- Arm 2- Hypothyroid treatment naïve patients: The subjects will be identified and selected from clinical settings such as hospitals, clinics and certified laboratories.

INTERVENTIONS:
Diagnostic Test: Blood test for Thyroid stimulating hormone (TSH) — Blood test for Thyroid stimulating hormone (TSH)
  Groups: Arm 1-Healthy Volunteers

SUMMARY:
Type of Study Questionnaire- Development and validation

Information about the Q'SHY:

* The Q'SHY- Questionnaire for Screening of Hypothyroidism is a Patient Reported Outcome (PRO) tool to enable screening for Hypothyroidism in the general population.
* It is a 20-item questionnaire which covers aspects of the symptoms of Hypothyroidism and incorporates the contributory factors from patient history which when combined, provides a robust tool to effectively screen the population.
* The questionnaire content is being created based on a thorough search for relevant literature and encompasses all important aspects for screening purposes

DETAILED DESCRIPTION:
Objectives The objectives of the study are as described in the below points.

1. To develop a questionnaire (Q'SHY) for the identification and screening of subjects with suspected hypothyroidism.
2. To assess the validity of the designed questionnaire by comparing the outcomes of the responses between General population subjects and treatment naïve subjects group with hypothyroidism.
3. The study aims to establish a valid questionnaire with a robust sensitivity and specificity to detect signs and symptoms of hypothyroidism.

Inclusion criteria for Subjects The criteria based on which, subjects in each Arm will be chosen to take part in the survey. Arm1: Subjects from the general population who are naïve to their hypothyroid status.

* Male and female subjects between the age of 18 years and 65 years
* Willing to sign the Subject Authorization Form (SAF) Arm 2: Subjects who are newly diagnosed patients of Hypothyroidism and are treatment naïve*.
* Male and female subjects between the ages 18 years and 65 years.
* Subjects who had symptoms of hypothyroidism were seen by a physician and diagnosed with hypothyroidism after laboratory testing of Thyroid Stimulating Hormone > 4.5 Milli international units per litre(mIU/L) within 2 weeks from the date of the survey
* Willing to sign the SAF
* Willing to provide their Thyroid Function Test report that was used to diagnose Hypothyroidism. * Treatment naive diagnosed on basis lab and clinical diagnosis within last 2 weeks

Exclusion criteria for subjects Arm 1: Subjects from the general population who are naïve to their hypothyroid status

* Individuals less than 18 years of age and more than 65 years of age.
* Pregnant or lactating females Subjects previously diagnosed with and received treatment for thyroid diseases.
* Subjects not willing to sign the SAF.

Arm 2: Subjects who are newly diagnosed patients of Hypothyroidism and are treatment naïve

* Individuals less than 18 years of age and more than 65 years of age.
* Pregnant or lactating females
* Subjects previously diagnosed with and received treatment for thyroid diseases.
* Patients on treatment for Thyroid diseases Subjects not willing to sign the SAF.

The above-mentioned criteria will be applicable to both Face validation and Pilot survey.

1. Subjects are divided into 2 arms, with 100 subjects in each arm.
2. Phase -1

   * Arm 1: Sixteen subjects from the general population who are naïve to their hypothyroid status with equal distribution of males and females.
   * Arm 2: Sixteen subjects who are newly diagnosed patients of Hypothyroidism are treatment naïve with equal distribution of males and females
3. Phase -2

   * Arm 1: One hundred subjects from the general population who are naïve to their hypothyroid status with equal distribution of males and females
   * Arm 2: One hundred subjects who are newly diagnosed patients of Hypothyroidism are treatment naïve with equal distribution of males and females

ELIGIBILITY:
Inclusion Criteria:

* The criteria based on which, subjects in each Arm will be chosen to take part in the survey. Arm 1: Subjects from the general population who are naïve to their hypothyroid status.

  * Male and female subjects between the age of 18 years and 65 years
  * Willing to sign the Subject Authorization Form (SAF) Arm 2: Subjects who are newly diagnosed patients of Hypothyroidism and are treatment naïve*.
  * Male and female subjects between the ages 18 years and 65 years.
  * Subjects who had symptoms of hypothyroidism, were seen by a physician and diagnosed with hypothyroidism after laboratory testing of TSH > 4.5 mIU/L within 2 weeks from the date of survey
  * Willing to sign the SAF
  * Willing to provide their Thyroid Function Test report that was used to diagnose Hypothyroidism. * Treatment naive diagnosed on basis lab and clinical diagnosis within last 2 weeks

Exclusion Criteria:

* Arm 1: Subjects from the general population who are naïve to their hypothyroid status

  * Individuals less than 18 years of age and more than 65 years of age.
  * Pregnant or lactating females
  * Subjects previously diagnosed with and received treatment for thyroid diseases.
  * Subjects not willing to sign the SAF. Arm 2: Subjects who are newly diagnosed patients of Hypothyroidism and are treatment naïve
  * Individuals less than 18 years of age and more than 65 years of age.
  * Pregnant or lactating females
  * Subjects previously diagnosed with and received treatment for thyroid diseases.
  * Patients on treatment for Thyroid diseases Subjects not willing to sign the SAF.

The above-mentioned criteria will be applicable to both Face validation and Pilot survey.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Phase -1
  * Arm 1: Sixteen subjects from the general population who are naïve to their hypothyroid status with equal distribution of males and females.
  * Arm 2: Sixteen subjects who are newly diagnosed patients of Hypothyroidism are treatment naïve with equal distribution of males and females
  Phase -2
  * Arm 1: One hundred subjects from the general population who are naïve to their hypothyroid status with equal distribution of males and females
  * Arm 2: One hundred subjects who are newly diagnosed patients of Hypothyroidism are treatment naïve with equal distribution of males and females
Sampling Method: Non-Probability Sample
Enrollment: 232 (Estimated)
Dates: Start 2021-01-18 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
To be able to develop a questionnaire (Q'SHY) for the identification and screening of subjects with suspected hypothyroidism | through out the study upto 1 year
  The aim is to develop a questionnaire considering literature review for symptoms selection, medical review of symptoms appropriateness, assigning weightage & questionnaire construction followed by expert review to construct a questionnaire
To be able to assess the validity of the designed questionnaire by comparing the outcomes of the responses between General population subjects and treatment naïve subjects group with hypothyroidism. | through out the study upto 1 year
  Through this study, we want to assess the validity of the questionnaire after receiving and comparing responses received from healthy volunteers and treatment naïve subjects with hypothyroidism through out the study we will have face validation of survey questionnaire - Face validation of survey questionnaire in hypothyroidism naïve and treatment naïve patients of hypothyroidism, revision of questionnaire if required after expert review of validation results
To be able to establish a valid questionnaire with a robust sensitivity and specificity to detect signs and symptoms of hypothyroidism | through out the study upto 1 year
  in this, Pilot survey in hypothyroidism naïve and treatment naïve patients of hypothyroidism will be conducted and data will be analyzed and used to establish validation.

CONTACTS AND LOCATIONS:
Overall Officials: Shivani Acharya, Study Director — Abbott
Locations (11):
- India (11):
  - Diabecare, Mumbai, Maharashtra
  - Center for Diabetes and Endocrine care, Bangalore
  - Apollo Excelcare Hospital, Guwahati
  - Care Outpatient Centre, Hyderabad
  - FS Endocrine and Diabetic Centre, Hyderabad
  - Dr. MV Rama Mohan, MD, DM, Hyderabad
  - Diabetes Thyroid Endocrine Center, Jaipur
  - Healthy Lifestyle Clinic, Kolkata
  - Ananda Clinic, Kolkata
  - Khandelwal Diabetes Thyroid & Endocrinology Clinic, New Delhi
  - Chellaram Diabetes Institute, Pune

IPD SHARING:
Plan to Share IPD: No